CLINICAL TRIAL: NCT05482178
Title: The Potential Role of Resistance Exercise on Inflammasome Activation and Cytokines Levels in Obese Subjects
Brief Title: The Association of Resistance Exercise With the Inflammasome Activation in Obesity Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elisa Barron-Cabrera (Other)
Responsible Party: Sponsor-Investigator, Elisa Barron-Cabrera, Professor, Universidad Autónoma de Sinaloa
Organization: Universidad Autónoma de Sinaloa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE-FCNYG-2022-FEB-001
Record Dates: First submitted 2022-07-27; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Physical Activity; Resistance Exercise; Inflammation; Obesity
Keywords: Resistance training; inflammasome; Obesity
MeSH Terms: conditions — Motor Activity; Inflammation; Obesity

STUDY DESIGN:
Intervention Model Description: Experimental
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance exercise training plus hypocaloric diet (Experimental): The participants received a caloric restriction of 20% of total energy estimated with Mifflin formula plus a structured, planned, and controlled resistance exercise program by a personal trained. The participant received the exercise program instructions every week and they performed by the own, and record the heart rate of each session on a paper format. All the appointment were once a month by trained nutritionists, and all the participants received a nutritional recommendation for the obesity management and a balanced food plan.
  Interventions: Behavioral: Resistance exercise training plus hypocaloric diet
- Hypocaloric diet (Active Comparator): The participants received a caloric restriction of 20% of total energy estimated with Mifflin formula. All the appointment were once a month by trained nutritionists, and all the subjects received a nutritional recommendation for the obesity management and a balanced food plan.
  Interventions: Behavioral: Hypocaloric diet

INTERVENTIONS:
Behavioral: Resistance exercise training plus hypocaloric diet — The exercise program included 3 phases of progressive intervention: 1) Adaptation which included 3-4 days per week at 60% of maximum heart rate, 2) Development phase which included 5 days per week at 75-85% of maximum heart rate and the last one, 3) Maintenance phase which included 5 days per week at 75-90% of maximum heart rate. The control and follow up will be through text message exchanges at least once a week or as many as necessary.
  On the other hand, the diet intervention consisted a caloric restriction of 20% of total energy estimated with Mifflin formula. The nutrients distributions are 50% for carbohydrates, 20% for protein and 30% for lipids, ensuring a sufficient intake of fiber (>25g per day).
  Arms: Resistance exercise training plus hypocaloric diet
Behavioral: Hypocaloric diet — The diet intervention consisted a caloric restriction of 20% of total energy estimated with Mifflin formula. The nutrients distributions are 50% for carbohydrates, 20% for protein and 30% for lipids, ensuring a sufficient intake of fiber (>25g per day).
  Arms: Hypocaloric diet

SUMMARY:
The intervention study consist in 3 months of follow up to evaluate the effect of resistance exercise on NLRP3 and interleukin-18 (IL-18) gene expression, and IL-18 and IL-1b cytokines levels in obese subjects, due to, the current evidence has been suggested that aerobic physical exercise could reduce the low-grade chronic inflammation through the downregulation of the NLRP3 inflammasome in obesity subjects, however, there are not enough evidence with resistance protocol. The investigator randomized into two intervention groups: a) group with resistance exercise training plus hypocaloric diet, and b) group with hypocaloric diet. The blood sample was taken fasting at baseline and final intervention (3rd month). The serum was separated for biochemical analyzes and the quantification of cytokines levels. The RNA was obtained from leukocytes to expression assay.

DETAILED DESCRIPTION:
Obesity is a metabolic condition with a high worldwide prevalence. It is characterized by low-grade chronic inflammation and high cytokines level as consequence of the excessive accumulation of adipose tissue. The NLRP3 protein is part of the NLRP3 inflammasome, a multiprotein complex related to inflammation and the risk of developing metabolic disorders. In this sense, the evidence has been suggested that physical exercise could reduce the inflammation through the downregulation of the NLRP3 inflammasome. The aim of this study is evaluate the effect of resistance exercise on NLRP3 and IL-18 gene expression and and IL-18 and IL-1b cytokines levels in obese subjects. This is an experimental study with 3 months of follow up. Participants were randomized into two intervention groups: a) group with resistance exercise plus hypocaloric diet, and b) group with hypocaloric diet. The exercise program was design by certified personal trained, and consisted in 3 phases: conditioning, development and maintenance. Dietary information was collect by validated retrospective questionnaires (24-hour record and 3-days dietary diary) and analyzed in Nutritionist Pro software. Body composition was evaluated by bioimpedance. The biochemical analyzes were performed on serum sample using spectrophotometry equipment. RNA was obtained from leukocytes from peripheral blood, cDNA synthesis was performed with a ThermoFisher kit, and the expression assay was performed by real-time polymerase chain reaction (PCR) using Taqman probes with the 2-ΔΔcq relative quantification method. Cytokines quantification were perform using a commercial ELISA kit. Statistical analysis will be using the Statistical Package for Social Sciences (SPSS v.25) software and a value of p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Both sex
* Older than 25 years old
* Women with waist circumference ≥ 80cm and men with ≥ 90cm
* Subjects with BMI between 30 and 40 kg/m2

Exclusion Criteria:

* Subjects with diagnosis of metabolic alterations
* Subjects with chronic pharmacological treatment
* Subjects with anti-inflammatories drugs prescription

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-12-16 (Estimated)

PRIMARY OUTCOMES:
NLRP3 gene expression | Change from baseline NLRP3 gene expression at 3 months
  Assay expression will be performed by real-time PCR using Taqman probes with the 2-ΔΔcq relative quantification method
IL-18 gene expression | Change from baseline IL-18 gene expression at 3 months
  Assay expression will be performed by real-time PCR using Taqman probes with the 2-ΔΔcq relative quantification method
IL-18 cytokine | Change from baseline IL-18 cytokine at 3 months
  commercial ELISA kit
IL-1b cytokine | Change from baseline IL-1b cytokine at 3 months
  commercial ELISA kit

SECONDARY OUTCOMES:
Weight | Change from baseline weight at 3 months
  Weighing machine using bioimpedance technology
Body fat mass | Change from baseline body fat mass at 3 months
  Weighing machine using bioimpedance technology
Serum triglycerides | Change from baseline serum triglycerides at 3 months
  Liquid chemistry using spectrum equipment
Serum cholesterol | Change from baseline serum cholesterol at 3 months
  Liquid chemistry using spectrum equipment
Serum glucose | Change from baseline serum glucose at 3 months
  Liquid chemistry using spectrum equipment

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Barron, PhD, Principal Investigator — Autonomous University of Sinaloa
Locations (1):
- Autonomous University of Sinaloa, Culiacán, Sinaloa, Mexico

IPD SHARING:
Plan to Share IPD: No
We reserve to respect the individual rights of not revealing personal data of the participants, since this information is signing in the informed consent. However, we will publish all the results on a manuscript.

REFERENCES:
- [Background] Metsios GS, Moe RH, Kitas GD. Exercise and inflammation. Best Pract Res Clin Rheumatol. 2020 Apr;34(2):101504. doi: 10.1016/j.berh.2020.101504. Epub 2020 Apr 2. PMID 32249021
- [Background] Izaola O, de Luis D, Sajoux I, Domingo JC, Vidal M. [Inflammation and obesity (lipoinflammation)]. Nutr Hosp. 2015 Jun 1;31(6):2352-8. doi: 10.3305/nh.2015.31.6.8829. Spanish. PMID 26040339
- [Background] Ozaki E, Campbell M, Doyle SL. Targeting the NLRP3 inflammasome in chronic inflammatory diseases: current perspectives. J Inflamm Res. 2015 Jan 16;8:15-27. doi: 10.2147/JIR.S51250. eCollection 2015. PMID 25653548
- [Background] You T, Berman DM, Ryan AS, Nicklas BJ. Effects of hypocaloric diet and exercise training on inflammation and adipocyte lipolysis in obese postmenopausal women. J Clin Endocrinol Metab. 2004 Apr;89(4):1739-46. doi: 10.1210/jc.2003-031310. PMID 15070939
- [Result] Barron-Cabrera E, Gonzalez-Becerra K, Rosales-Chavez G, Mora-Jimenez A, Hernandez-Canaveral I, Martinez-Lopez E. Low-grade chronic inflammation is attenuated by exercise training in obese adults through down-regulation of ASC gene in peripheral blood: a pilot study. Genes Nutr. 2020 Aug 27;15(1):15. doi: 10.1186/s12263-020-00674-0. PMID 32854610
- [Result] Butts B, Butler J, Dunbar SB, Corwin E, Gary RA. Effects of Exercise on ASC Methylation and IL-1 Cytokines in Heart Failure. Med Sci Sports Exerc. 2018 Sep;50(9):1757-1766. doi: 10.1249/MSS.0000000000001641. PMID 29683921
- [Result] Nakajima K, Takeoka M, Mori M, Hashimoto S, Sakurai A, Nose H, Higuchi K, Itano N, Shiohara M, Oh T, Taniguchi S. Exercise effects on methylation of ASC gene. Int J Sports Med. 2010 Sep;31(9):671-5. doi: 10.1055/s-0029-1246140. Epub 2010 Mar 3. PMID 20200803